CLINICAL TRIAL: NCT02896543
Title: The Relationship of Change of Dendritic Cells Fractalkine and P-selectin in Patients With Acute Myocardial Infarction
Brief Title: The Relationship of Change of Dendritic Cells Fractalkine and P-selectin Patients With Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Rchuang, Professor, The First Affiliated Hospital of Dalian Medical University
Other Study IDs: LCKY2016-6
Record Dates: First submitted 2016-07-06; First posted 2016-09-12 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Acute Myocardial Infarction
Keywords: dendritic cells; P-selectin
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- STEMI group: The study population consists of 30 patients with ST-elevated acute myocardial infarction (STEMI,n = 30) who are admitted within 24 hours after chest pain attacks. They will all undergo coronary angiography.The diagnosis is made according to American Heart Association (AHA, 2014 and 2015) guidelines. Patients who had obvious blood system diseases,severe liver dysfunction, severe renal insufficiency,severe heart failure (NYHA class 3 and 4), acute or chronic infectious diseases, disease of immune system, asthma, malignant tumor, other advanced disease are excluded.
  Interventions: Other: measurement
- Control group: 15 age and body mass index matched healthy subjects with neither coronary artery disease nor any of the components of the metabolic syndrome are enrolled as Control group.
  Interventions: Other: measurement

INTERVENTIONS:
Other: measurement — Blood is obtained into ethylene diamine tetraacetic acid（EDTA） tubes from all subjects via antecubital vein puncture to measure the number of dendritic cells(DCs) and the concentration of sP-selectin. The number of dendritic cells(DCs) and the concentration of sP-selectin are measured in all patients with STEMI at 0 and 5-7 days after admission. The number of dendritic cells(DCs) and the only once in control group after admission.

SUMMARY:
This study evaluates the relationship of change of dendritic cells fractalkine and P-selectin in patients with acute myocardial infarction.

DETAILED DESCRIPTION:
Dendritic cells (DCs) are the most potent antigen-presenting cells, with the unique ability to initiate a primary immune response to certain antigens by activation of "naive" T cells, and are actively related to the process of atherosclerosis. Two DC subsets, myeloid DCs (mDCs) and plasmacytoid DCs (pDCs), were identified in humans. In our previous study, the investigators found that change of dendritic cells and fractalkine in patients with acute myocardial infarction. At the same time, the level of P-selectin increased. In addition, the interaction of dendritic cells and P-selectin promotes the progress of atherosclerosis. In this study, the investigators want to see whether the balance between mDCs and pDCs is altered in patients with acute myocardial infarction. sP-selectin is one of the members of the family of proteins, mediate leukocyte adhesion and rolling in vascular endothelial, studies have shown that in patients with unstable angina and acute myocardial infarction in serum sP-selectin protein increased significantly, showed that sP-selectin associated with the activity of coronary heart disease, causing plaque instability.However, there is few relevant studies about the relationship of dendritic cells and P-selectin in patients with acute myocardial infarction. This study valuates the relationship of dendritic cells and P-selectin in patients with acute myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as STEMI.
* with left ventricular ejection fraction（LVEF）>=45%
* written informed consents are obtained.
* admitted within 24 hours after chest pain attacked.

Exclusion Criteria:

* Obvious blood system diseases.
* Combination with other organs function failure: severe liver dysfunction, severe renal insufficiency,severe heart failure (NYHA class 3 and 4), acute or chronic infectious diseases, disease of immune system, asthma, malignant tumor, other advanced disease, etc.
* Pregnant women and planned pregnancy women.
* With drug allergy or contraindications.
* refusal to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with STEMI.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The number of dendritic cells(DCs)(percentage of total white blood cells) and the concentration of sP-selectin(ng/ml) within 24 hours after chest pain attacks | 24 hours
  The number of dendritic cells(DCs) in percentage of total white blood cells;the concentration of sP-selectin in ng/ml

SECONDARY OUTCOMES:
Change of peripheral blood DCs number (percentage of total white blood cells) and its fractalkine change of peripheral blood DCs number(percentage of total white blood cells) within 1 week after chest pain attacks | 1 week
  Dendritic cells(DCs) number in percentage of total white blood cells;its fractalkine change of peripheral blood DCs in percentage of total white blood cells

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laszik Z, Jansen PJ, Cummings RD, Tedder TF, McEver RP, Moore KL. P-selectin glycoprotein ligand-1 is broadly expressed in cells of myeloid, lymphoid, and dendritic lineage and in some nonhematopoietic cells. Blood. 1996 Oct 15;88(8):3010-21. PMID 8874199
- [Result] Hussain M, Javeed A, Ashraf M, Riaz A, Mushtaq MH. Aspirin may do wonders by the induction of immunological self-tolerance against autoimmune atherosclerosis. Med Hypotheses. 2012 Jan;78(1):171-3. doi: 10.1016/j.mehy.2011.10.019. Epub 2011 Nov 8. PMID 22070887
- [Result] Packard RR, Lichtman AH, Libby P. Innate and adaptive immunity in atherosclerosis. Semin Immunopathol. 2009 Jun;31(1):5-22. doi: 10.1007/s00281-009-0153-8. Epub 2009 May 16. PMID 19449008
- [Result] Kieffer JD, Fuhlbrigge RC, Armerding D, Robert C, Ferenczi K, Camphausen RT, Kupper TS. Neutrophils, monocytes, and dendritic cells express the same specialized form of PSGL-1 as do skin-homing memory T cells: cutaneous lymphocyte antigen. Biochem Biophys Res Commun. 2001 Jul 20;285(3):577-87. doi: 10.1006/bbrc.2001.5230. PMID 11453631
- [Result] Schakel K, Kannagi R, Kniep B, Goto Y, Mitsuoka C, Zwirner J, Soruri A, von Kietzell M, Rieber E. 6-Sulfo LacNAc, a novel carbohydrate modification of PSGL-1, defines an inflammatory type of human dendritic cells. Immunity. 2002 Sep;17(3):289-301. doi: 10.1016/s1074-7613(02)00393-x. PMID 12354382
- [Result] Bonasio R, Scimone ML, Schaerli P, Grabie N, Lichtman AH, von Andrian UH. Clonal deletion of thymocytes by circulating dendritic cells homing to the thymus. Nat Immunol. 2006 Oct;7(10):1092-100. doi: 10.1038/ni1385. Epub 2006 Sep 3. PMID 16951687
- [Result] Yao K, Lu H, Huang R, Zhang S, Hong X, Shi H, Sun A, Qian J, Zou Y, Ge J. Changes of dendritic cells and fractalkine in type 2 diabetic patients with unstable angina pectoris: a preliminary report. Cardiovasc Diabetol. 2011 Jun 10;10:50. doi: 10.1186/1475-2840-10-50. PMID 21658276